CLINICAL TRIAL: NCT03450967
Title: A Phase II Study of Durvalumab (MEDI4736) Plus Tremelimumab Combined With Proton Therapy for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Durvalumab Plus Tremelimumab Combined With Proton Therapy for HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-09-026
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab Plus Tremelimumab (Experimental): Durvalumab 1500mg plus tremelimumab 75mg via IV infusion Q4W, starting on Week 0, for up to a maximum of 4 doses/cycles followed by durvalumab monotherapy 1500mg via IV infusion Q4W, starting 4 weeks after the last infusion of the combination until progression.).
  Interventions: Drug: Durvalumab Plus Tremelimumab

INTERVENTIONS:
Drug: Durvalumab Plus Tremelimumab — Durvalumab 1500mg plus tremelimumab 75mg via IV infusion Q4W, starting on Week 0, for up to a maximum of 4 doses/cycles followed by durvalumab monotherapy 1500mg via IV infusion Q4W, starting 4 weeks after the last infusion of the combination until progression.).

SUMMARY:
* Clinical Phase: phase II single arm study
* Primary Objectives: Response rate
* Number of Subjects: 27 patients
* Study Population: recurrent or metastatic head and neck squamous cell carcinoma
* Investigational Product(s), Dose, and Mode of Administration:

Durvalumab 1500mg plus tremelimumab 75mg via IV infusion Q4W, starting on Week 0, for up to a maximum of 4 doses/cycles followed by durvalumab monotherapy 1500mg via IV infusion Q4W, starting 4 weeks after the last infusion of the combination until progression.).

Proton therapy 5 GyE x 5 fractions

- Study Assessments and Criteria for Evaluation: Safety Assessments: according to NCI CTCAE version 4.0 Efficacy Assessments: according to RECIST version 1.1

- Statistical Methods and Data Analysis: PFS: from the date of treatment to the date of progression or death or last follow-up OS: from the date of treatment to the date of death or last follow-up

- Sample Size Determination: Patients must have a histologically confirmed diagnosis of HNSCC. In this phase II study, up to approximately 27 eligible patients will be enrolled. It is anticipated that full accrual to this study will take approximately 24 months.

H0: Objective response rate ≤10% H1: Objective response rate ≥35% According to Simon's two-stage optimal design (power of 90% and one-sided alpha of 0.05), this study needs total 27 evaluable patients. At the first stage, 11 patients would be enrolled. If two or more among them achieve objective response, the study will go forward the second stage. At the second stage, 16 additional patients (total 27 patients) would be enrolled. Among the total 27 evaluable patients, six or more objective responses are necessary for this drug to be evaluated further in the group of R/M HNSCC

DETAILED DESCRIPTION:
The incidence of Head and neck cancer (HNC) is approximately 6% of all cases with a world annual incidence and nearly 90 to 95% of HNC is squamous cell carcinoma (HNSCC). [1] For patients with recurrent or metastatic HNSCC (R/M HNSCC), cytotoxic-based chemotherapy remains the standard therapeutic option. The median survival of these patients treated with cytotoxic-based chemotherapy, however, is only 6 to 10 months. For those who are not candidates for chemotherapy, the prognosis is even worse with median survival of 3 to 6 months. [2-4] Thus, new therapeutic options for these patients are needed to improve the treatment outcomes.

We hypothesize that durvalumab plus tremelimumab combined with proton therapy would be effective in R/M HNSCC.

The combination of immunotherapy and RT can be effective regimen because immunologic response might be enhanced by RT through the alteration of microenvironment within the irradiated field, tumor antigen release and "abscopal effect" at distant metastatic sites. In addition, the benefit of proton therapy is to deliver RT dose just to target lesion. The irradiated volume can be significantly reduced with proton therapy compared to X-ray treatment, thus proton therapy will provide better quality of life compared to X-ray during palliative RT.

Patients in the durvalumab (MEDI4736) + tremelimumab combination therapy treatment group will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) for up to 4 doses/cycles each, followed by durvalumab (MEDI4736) 1500mg Q4W until confirmed disease progression unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. The first durvalumab (MEDI4736) monotherapy dose at 1500mg Q4W will be 4 weeks after the final dose of durvalumab (MEDI4736) in combination with tremelimumab.

Tremelimumab will be administered first; the durvalumab (MEDI4736) infusion will start approximately 1 hour (maximum 2 hours) after the end of the tremelimumab infusion. If there are no clinically significant concerns after the first cycle, then, at the discretion of the Investigator, all other cycles of durvalumab (MEDI4736) can be given immediately after the tremelimumab infusion has finished.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven HNSCC

  * Inoperable or metastatic disease

    * Age ≥18years

      * More than one previous chemotherapy including at least one platinum-based regimen

        * ECOG performance status of 0 to 1

          * At least two measurable lesions

            ⑦ Adequate organ function as evidenced by the following; Haemoglobin ≥ 9.0 g/dl Absolute neutrophil count (ANC) > 1.0 x 109/L platelets > 100 x 109/L serum bilirubin ≤1.5 institutional upper limit of normal (ULN); AST(SGOT) and/or ALT(SGPT) ≤ 2.5 x ULN unless liver metastases are present, in which case it must be ≤ 5 x ULN creatinine clearance ≥ 40mL/min by Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance

            ⑧ Body weight > 30kg

            ⑨ Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy). Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause

            ⑩ Written informed consent form

            ⑪ Patients who could submit at least one unstained slide to evaluate the PD-L1 expression status (PD-L1 status, which is positive (expression > 1% of tumor cells) or negative, is the prerequisite for the enrollment. If the submitted slides are unacceptable for the analysis for PD-L1 and there is no remained slide, the patient cannot be enrolled)

            ⑫ Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
2. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) ≤ 30 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca and the investigator
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

   Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
4. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
5. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
6. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
7. History of allogenic organ transplantation.
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   Patients with vitiligo or alopecia Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement Any chronic skin condition that does not require systemic therapy Patients without active disease in the last 5 years may be included but only after consultation with the study physician Patients with celiac disease controlled by diet alone
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
10. History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in situ without evidence of disease
11. History of leptomeningeal carcinomatosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Response rate | about 24months
  according to RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided